CLINICAL TRIAL: NCT03859089
Title: Cannabis for Opioid Substitution Trial
Acronym: COST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cannabis Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: 17-96275KCRA
Record Dates: First submitted 2017-07-22; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Pain Syndrome; Opioid Use; Cannabis Use
Keywords: medical cannabis; opioids; pain; substitution; alternative
MeSH Terms: conditions — Somatoform Disorders; Pain | interventions — Medical Marijuana

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Medical Cannabis — N/A - Observational Cohort Study

SUMMARY:
The purpose of this study is to define common strains of cannabis that adult chronic cancer and non-cancer pain syndrome patients are using as a replacement for opioids (narcotics). Identified strains, if any, will then be tested via randomized controlled trials to support an application for a Health Canada Drug Identification Number.

DETAILED DESCRIPTION:
The search for safer alternatives to opioids for treating chronic cancer and non-cancer pain syndromes currently is an important initiative. Cannabis Research Associates (CRA) has been commissioned by Northern Green Canada Inc. to conduct a multi-phase study that will first define common strains of cannabis that patients use as a replacement for opioids, then conduct a randomized controlled trial to support an application to Health Canada for a Drug Identification Number. This protocol summarizes the methods for phase I.

In total, the Investigators plan to recruit 1,200 adult patients (> 25 years) currently using cannabis to treat chronic cancer and non-cancer pain syndromes conditions. Patients will be recruited from six pain clinics throughout Ontario. Pain clinics have not yet been identified. The study Investigators will invite licensed physicians from various private pain clinics to collaborate on this study.

This is an observational cohort study involving a mixed methods approach. Patients interested in participating will have the option to have an online survey link emailed to them so they can complete the survey at a convenient time. Or, patients can choose to complete the online survey in person with the assistance of a Research Assistant. Research Assistants will have hard copy surveys to serve as a back-up solution should they be faced with Internet connectivity and/or online survey hosting issues. No personal identifying information will be collected. Hard copy data will be stored in locked cabinets and shipped via courier to Cannabis Research Associates in batches.

All aspects of this study will be executed under the supervision of the study Investigators. Scientific independence from the sponsoring body will be maintained, and no censorship of data management, analysis, or presentation/publication will be permitted.

This study will be executed under the approval and ongoing supervision of the Research Ethics Board, as required.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients aged > 25 years-CPSO Policy states that physicians cannot prescribe medical cannabis to persons under the age of 25 unless all other conventional therapies have failed. Furthermore, there is evidence to support that cannabis use in younger persons can have lasting effects since the brain is still developing (Wier K, 2015).
2. English-speaking, or with the assistance of a family member/friend that can interpret English for the patient.
3. Qualifying medical diagnosis for appropriate use of medical cannabis by a licensed physician.
4. Current medical cannabis use to treat chronic cancer and non-cancer pain syndromes.
5. Current or past use of prescription opioids to treat chronic cancer and non-cancer pain syndromes.

Exclusion Criteria:

1. Patients taking medical cannabis for reasons other than chronic cancer and non-cancer pain syndromes

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic cancer and non-cancer pain syndrome patients currently taking medical cannabis and are currently or have previously taken opioids to treat pain.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-10-10 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Cannabis as replacement for opioids | Through study completion, an average of 1 year
  Define common strains of cannabis that patients are using as a replacement for opioids (should any exist)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Price, MD, Principal Investigator — Cannabis Research Associates
Locations (1):
- Synergy Health Services Inc., Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
N/A - no plans to share individual participant data.